CLINICAL TRIAL: NCT07129421
Title: A Prospective, Randomized, Multicenter Evaluation of the Safety and Effectiveness of the EMBLOK™ Embolic Protection System Compared With No Cerebral Embolic Protection During Transcatheter Aortic Valve Replacement
Brief Title: Evaluation of Safety and Effectiveness of the EMBLOK EPS Compared With No Cerebral Embolic Protection During TAVR
Acronym: EMBLOK II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emblok, Inc. (Industry)
Collaborators: Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLP 002-2025
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: AORTIC VALVE DISEASES; Aortic Valve Stenosis and/or Insufficiency; Aortic Valve Regurgitation; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Parallel Assignment This prospective, multicenter, single-blind, randomized controlled trial will enroll up to a total of 560 subjects undergoing TAVR at up to 40 investigational sites in the United States.
  Prior to enrollment of the first randomized subject at each site, each site will enroll 2 Roll-In subjects (up to 80 subjects total), who will not be randomized but will receive the EMBLOK EPS during TAVR.
  In the randomized cohort, up to 480 subjects meeting eligibility criteria will be randomized 1:1 (stratified by operative risk and study site) to one of two treatment arms:
  Intervention - EMBLOK EPS during TAVR Control - Unprotected TAVR
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. The following individuals will be blinded to the subject's treatment allocation:
  Site personnel administering neurological evaluations DW-MRI Core Laboratory personnel performing imaging analyses
  While subjects and their family members will not be blinded, they should not be explicitly informed of their treatment group assignment to minimize the risk of inadvertent unblinding of site personnel administering neurological evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- EMBLOK™ Embolic Protection System (Experimental): Device Description:
  The EMBLOK™ Embolic Protection System ("EMBLOK EPS") is a sterile, single use system designed to capture and remove debris (e.g., thrombus, calcium, atheroma) dislodged during transcatheter aortic valve replacement (TAVR) procedures. The device is currently for investigational use only.
  When Device Will Be Used:
  Roll-in: Prior to enrollment of the first randomized subject at each site, each site will enroll 2 Roll-In subjects, who will not be randomized but will receive the EMBLOK EPS during TAVR.
  Randomized: Up to 480 subjects meeting eligibility criteria will be randomized 1:1. The experimental "intervention" arm is utilizing EMBLOK EPS during TAVR (up to 240 subjects).
  Interventions: Device: EMBLOK™ Embolic Protection System ("EMBLOK EPS")
- Unprotected TAVR (No Intervention): The control comparator is TAVR without the use of a cerebral embolic protection device ("unprotected TAVR").

INTERVENTIONS:
Device: EMBLOK™ Embolic Protection System ("EMBLOK EPS") — The EMBLOK EPS is intended to capture and remove thrombus/debris while performing transcatheter aortic valve replacement procedures.
  Arms: EMBLOK™ Embolic Protection System

SUMMARY:
The objective of the study is to evaluate the safety, effectiveness, and performance of the EMBLOK EPS during TAVR by randomized comparison with TAVR without embolic protection (unprotected TAVR). The targeted study population consists of patients meeting FDA-approved indications for TAVR with commercially available transcatheter heart valve systems.

This prospective, multicenter, single-blind, randomized controlled trial will enroll up to a total of 560 subjects undergoing TAVR at up to 40 investigational sites in the United States. All subjects will undergo clinical follow-up (including detailed neurological assessments) in-hospital and at 30 days, and diffusion-weighted magnetic resonance imaging (DW-MRI) follow-up at 24 to 36 hours post-procedure.

DETAILED DESCRIPTION:
Embolic stroke remains a major complication for TAVR, resulting in a two-fold increase in 1-year mortality. Embolic protection devices have been developed to filter embolic debris during the procedure, potentially reducing the occurrence of neurologic events associated with TAVR. The EMBLOK EPS may improve on currently available devices by capturing and retrieving debris directed toward all 3 cerebral vessels in the aortic arch as well as the descending aorta.

The objective of the study is to evaluate the safety, effectiveness, and performance of the EMBLOK EPS during TAVR by randomized comparison with TAVR without embolic protection (unprotected TAVR).

The targeted study population consists of patients meeting FDA-approved indications for TAVR with commercially available transcatheter heart valve systems.

This prospective, multicenter, single-blind, randomized controlled trial will enroll up to a total of 560 subjects undergoing TAVR at up to 40 investigational sites in the United States.

Prior to enrollment of the first randomized subject at each site, each site will enroll 2 Roll-In subjects (up to 80 subjects total), who will not be randomized but will receive the EMBLOK EPS during TAVR.

In the randomized cohort, up to 480 subjects meeting eligibility criteria will be randomized 1:1 (stratified by operative risk and study site) to one of two treatment arms:

1. Intervention - EMBLOK EPS during TAVR
2. Control -Unprotected TAVR

All subjects will undergo clinical follow-up (including detailed neurological assessments) in-hospital and at 30 days, and diffusion-weighted magnetic resonance imaging (DW-MRI) follow-up at 24 to 36 hours post-procedure.

ELIGIBILITY:
Clinical Eligibility Criteria:

Clinical Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for participation in the study:

1. Subject is ≥ 18 years of age.
2. Subject meets FDA approved indications for TAVR using an iliofemoral approach with a commercially approved transcatheter heart valve.
3. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to the index study procedure.
4. Subject agrees to comply with all protocol-specified procedures and assessments.
5. Subject or subject's legal representative signs an IRB/EC approved informed consent form prior to study participation.

Clinical Exclusion Criteria:

Subjects will be excluded if any of the following criteria apply:

1. Subjects with hepatic failure (Child-Pugh class C).
2. Subjects with hypercoagulable states that cannot be corrected by additional periprocedural heparin.
3. Subjects who have a planned treatment with any other investigational device or procedure during the study period.
4. Subjects planned to undergo any other cardiac surgical or interventional procedure (e.g., concurrent coronary revascularization) during the TAVR procedure or within 10 days prior to the TAVR procedure. NOTE: Diagnostic cardiac catheterization is permitted within 10 days prior to the TAVR procedure.
5. Subject has experienced an acute myocardial infarction (World Health Organization [WHO] criteria) within 30 days of the planned index procedure.
6. Subject requires an urgent or emergent TAVR procedure.
7. Subjects with renal failure (estimated Glomerular Filtration Rate [eGFR] < 30 mL/min by the Modification of Diet in Renal Disease [MDRD] formula, or on dialysis).
8. Subject has documented history of stroke or transient ischemic attack within prior 6 months, or any prior stroke with a permanent major disability or deficit (baseline mRS ≥3).
9. Subject has an ejection fraction of 30% or less.
10. Subject has a sensitivity to contrast media that cannot be adequately pre-treated.
11. Subject has known allergy or hypersensitivity to any embolic protection device materials (e.g., nickel-titanium) or allergy to intravascular contrast agents that cannot be pre-medicated.
12. Subject has active endocarditis or an ongoing systemic infection defined as fever with temperature > 38°C and/ or white blood cell > 15,000 IU.
13. Subjects undergoing therapeutic thrombolysis.
14. Subject has history of bleeding diathesis or a coagulopathy or contraindications to anticoagulation and antiplatelet therapy.
15. Subject is known or suspected to be pregnant, or is lactating.
16. Subject has contraindications to cerebral MRI (e.g., body habitus that precludes imaging, claustrophobia, implanted non-MRI compatible permanent pacemaker or defibrillator, metallic clips or fragments).
17. In the investigator's opinion, the subject has other factors that may cause the subject to be non-compliant with the protocol or confound the data interpretation, such as participating in another drug or device clinical study, or other medical illness.

General Anatomic Exclusion Criteria

Subjects meeting any of the following criteria will not be eligible for participation in the study:

1. Non-iliofemoral approach is required for the TAVR system (e.g., trans-axillary, trans-subclavian, trans-brachiocephalic, trans-carotid, trans-apical or trans-aortic access for TAVR is required).
2. Subject peripheral anatomy is not compatible with contralateral iliofemoral access with an 11 French catheter (e.g., due to excessive tortuosity, stenosis, ectasia, dissection, or aneurysm).
3. Ascending aorta length (from the brachiocephalic artery takeoff to the most distal edge of the TAVR prosthetic device) less than 3.5 cm.
4. Diameter of the aorta at the intended site of Emblok filter deployment proximal to the brachiocephalic artery ostium is less than 25 mm or greater than 40 mm.
5. Subjects with severe peripheral arterial, abdominal aortic, or thoracic aortic disease that precludes delivery sheath vascular access.
6. Subjects in whom the aortic arch is heavily calcified, severely atheromatous, or severely tortuous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-10-21 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | Evaluated at 72 hours post-procedure (TAVR)
  The primary efficacy endpoint is neuroprotection efficacy, determined by pair-wise comparisons among all subjects (Finkelstein-Schoenfeld [FS] method1) according to the following prespecified hierarchy of adverse outcomes:
  * Ischemic stroke (disabling or non-disabling) [evaluated at 72 hours post-procedure]
  * Total lesion volume by DW-MRI [evaluated at 24-36 hours post-procedure]
Primary Safety Endpoint | Evaluated at 30-day post-procedure (TAVR) follow-up visit
  The primary safety endpoint is Major Adverse Events, defined as the composite of the following components at 30 days:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Acute kidney injury (Stage 3)

SECONDARY OUTCOMES:
Combined Safety and Efficacy | Evaluated post-procedure (day 1), in-hospital (defined as 7 days post-procedure or immediately prior to discharge from the index procedure hospitalization, whichever occurs first)
  Combined safety and efficacy endpoint is defined as a composite of the following VARC-2 defined components, evaluated post-procedure and in-hospital:
  * All-cause mortality
  * All stroke (disabling and non-disabling) and transient ischemic attack (TIA)
  * Acute kidney injury - Stage 2 or 3 (including renal replacement therapy)
Mortality (VARC-2 defined) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up until 7 days post procedure, which ever occurs first.
  Mortality (VARC-2 defined), evaluated in-hospital, defined as All-cause mortality:
  * Cardiovascular mortality
  * Non-cardiovascular mortality
Neurological Events (VARC-2 and NeuroARC defined) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  Neurological Events (VARC-2 and NeuroARC defined)
  * Stroke (subclassified as ischemic, hemorrhagic, or undetermined, and as disabling or non-disabling)
  * TIA
Incidence of acute kidney injury (AKIN classification) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.]
  Incidence of acute kidney injury (AKIN classification), subclassified as stage 1, 2, or 3 Acute Kidney Injury (AKIN Classification)
  * AKI Stage 1
  * AKI Stage 2
  * AKI Stage 3
Incidence of major vascular complications (VARC-3 defined) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.]
  Vascular Complications
  • Major vascular complications
Incidence of life-threatening or disabling bleeding and major bleeding (VARC-2 defined) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  Bleeding Complications (VARC-2 defined)
  * Life-threatening or disabling bleeding
  * Major bleeding
Major adverse embolic events (MAEE) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up until 7 days post procedure, which ever occurs first.]
  Incidence of the composite of all stroke (disabling or non-disabling) and transient ischemic attack (TIA), and Acute Kidney Injury Stage 2 or 3 (including renal replacement therapy), and systemic embolization Major adverse embolic events (MAEE)
  MAEE will be reported as a composite and components [evaluated post-procedure and in-hospital]:
  * All stroke (disabling and non-disabling) or TIA
  * Acute kidney injury (Stage 2 or 3, including RRT)
  * Systemic embolization
Imaging Endpoints: Total volume of new post-procedure cerebral ischemic lesions | Evaluated 24-36 hours post-procedure
  Imaging Endpoints [assessed 24-36 hours post-procedure by an independent DW-MRI Core Laboratory]
  • Total volume of new post-procedure cerebral ischemic lesions (TLV) (reported as continuous and categorical measures)
Imaging Endpoints: Total supra-threshold cerebral ischemic lesion volume | Evaluated 24-36 hours post-procedure
  Imaging Endpoints [assessed 24-36 hours post-procedure by an independent DW-MRI Core Laboratory]
  • Total supra-threshold cerebral ischemic lesion volume (reported according to predefined thresholds)
Imaging Endpoints: Presence of new post-procedure cerebral ischemic lesions | Evaluated 24-36 hours post-procedure
  Imaging Endpoints [assessed 24-36 hours post-procedure by an independent DW-MRI Core Laboratory]
  • Presence of new post-procedure cerebral ischemic lesions
Imaging Endpoints: Number of new post-procedure cerebral ischemic lesions | Evaluated 24-36 hours post-procedure
  Imaging Endpoints [assessed 24-36 hours post-procedure by an independent DW-MRI Core Laboratory]
  • Number of new post-procedure cerebral ischemic lesions
Imaging Endpoints: Average new lesion volume | Evaluated 24-36 hours post-procedure
  Imaging Endpoints [assessed 24-36 hours post-procedure by an independent DW-MRI Core Laboratory]
  • Average new lesion volume
Imaging Endpoints: Largest per-subject single lesion | Evaluated 24-36 hours post-procedure
  Imaging Endpoints [assessed 24-36 hours post-procedure by an independent DW-MRI Core Laboratory]
  • Largest per-subject single lesion
Pathology Measures: Debris capture as the average number of captured particles ≥150 µm in diameter | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Pathology Measures [assessed post-procedure by an independent Pathology Core Laboratory only in subjects treated with EMBLOK EPS]
  • Debris capture, defined as the average number of captured particles ≥150 µm in diameter
Pathology Measures: Gross and histologic evaluation of captured debris | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Pathology Measures [assessed post-procedure by an independent Pathology Core Laboratory only in subjects treated with EMBLOK EPS]
  • Gross and histologic evaluation of captured embolic debris, including particle presence, count, size, and composition.
Neurocognitive Measures: NIHSS worsening | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.]
  Neurocognitive Measures
  • NIHSS worsening (increase of 2 or more from baseline)
Neurocognitive Measures: MoCA worsening | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.]
  Neurocognitive Measures
  • Montreal Cognitive Assessment (MoCA) worsening (decrease of 2 or more from baseline)
Secondary Device Performance Endpoints: Successful device deployment | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  • Successful device deployment, defined as ability to successfully deliver the device to the site of filter placement and successfully deploy the device.
Secondary Device Performance Endpoints: Successful device positioning | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  • Successful device positioning, defined as ability to position the device and to maintain the device in place for the duration of the TAVR procedure (as assessed by an independent Angiographic Core Laboratory)
Secondary Device Performance Endpoints: Successful device retrieval | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  • Successful device retrieval, defined as ability to retrieve the device intact
Secondary Device Performance Endpoints: Device success | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  • Device success, defined as successful deployment, positioning and retrieval
Secondary Device Performance Endpoints: Procedure success | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  • Procedure success, defined as device success in the absence of in-hospital embolic protection device-related major adverse cardiac and cerebrovascular events (MACCE). MACCE is defined as the composite of all-cause mortality, all stroke, and major vascular complications.

IPD SHARING:
Plan to Share IPD: No